CLINICAL TRIAL: NCT03786588
Title: Chronic Pelvic Pain With Vaginal Microbiota in Gestational Women Without HPV Infection
Brief Title: Patients With Chronic Pelvic Pain With Vaginal Microbiota
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, shuwang, Associate Professor, Peking Union Medical College Hospital
Other Study IDs: CPPVM
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Pelvic Pain
MeSH Terms: conditions — Pelvic Pain | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Vaginal microbiota in gestation CPP women without HPV infection
  Interventions: Other: Observation
- GroupB: Vaginal microbiota in gestation women without CPP and HPV infection

INTERVENTIONS:
Other: Observation — The patients with the negative results of HPV infection, and assigned to different group according to the CPP manifestation.
  Groups: Group A

SUMMARY:
Vaginal microorganisms play an important role in the occurrence and development of many diseases, such as persistent infection of high-risk human papillomavirus (HR-HPV) causing cervical intraepithelial neoplasia and cervical cancer, and the role of microorganisms in chronic prostatitis.

ELIGIBILITY:
Inclusion Criteria:

* Those are aged 20 to 45 years old, have vaginal intercourse more than 3 years, and aren't in menstrual, pregnancy or puerperium period.

Exclusion Criteria:

* Those are aged more than 45 years old without HPV infection in the last one year, having no vaginal intercourse, and those can't cooperate the examiner. Women who are HIV or hepatitis B/C positive, have autoimmune disorders and systemic disease (like diabetes mellitus, hormone treatment diseases, severe liver and kidney dysfunction), or have severe mental illness and malignant tumors are also excluded. At the same time, all the participants should meet the following requirements: no vagina douching within last 2 days, no vaginal intercourse within last 3 days, no systemic application of antifungal agents or antibiotics or pessaries within last 14 days of sampling.

Ages: 20 Years to 45 Years | Sex: Male
Age Groups: Adult
Study Population: Gestational participants without HPV infection
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2018-12-25 (Actual); Primary Completion 2019-12-25 (Estimated); Study Completion 2020-12-25 (Estimated)

PRIMARY OUTCOMES:
Vaginal microbiota difference | one year
  Vaginal microbiota difference between the women with or without CPP, and all the cases are cervical HPV negative.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China